CLINICAL TRIAL: NCT00941252
Title: Topical Imiquimod in Treating Patients With Grade 2/3 Cervical Intraepithelial Neoplasia
Brief Title: ITIC (Imiquimod Therapy in Cervical Intraepithelial Neoplasia)-Trial
Acronym: ITIC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof. MD. Paul Speiser, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITIC1.0
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imiquimod (Active Comparator): topical therapy for 16 weeks with imiquimod containing therapy
  Interventions: Drug: Topical imiquimod therapy
- Placebo (Placebo Comparator): topical therapy for 16 weeks with a placebo containing vaginal suppository
  Interventions: Drug: Topical imiquimod therapy

INTERVENTIONS:
Drug: Topical imiquimod therapy — therapy consists of treatment with topical vaginal suppositories for 16 weeks, each vaginal suppository contains 6.25mg of imiquimod, frequency (one time a week in treatment week 1+2, two times a week in treatment week 3+4, three times a week in treatment week 5-16)
  Other Names: Aldara

SUMMARY:
The present primary therapy of cervical intraepithelial neoplasia (CIN) grade 3 and persistent CIN 2 represents conisation. Surgical treatment can cause perioperative (infection, bleeding in in 5-10%) and postoperative (increased risk of preterm labor) complications, as well as incomplete resections (20%) and risk of recurrence in 5-17%. Imiquimod is an immunomodulating drug, that has been reported to be effective in human papilloma virus-related disease, such as vulvar intraepithelial neoplasia (VIN), vaginal intraepithelial neoplasia (VAIN), and anal intraepithelial neoplasia (AIN). The present randomised, placebo controlled, double blind study evaluates the efficacy of a topical treatment with imiquimod for 16 weeks in 60 patients with histologically confirmed CIN 2/3.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian women aged 18 years and older with proven HPV-associated CIN 2/3
* Colposcopy with fully visible transformation zone and lesion
* Safe Contraception
* Signed Informed Consent
* Negative urine pregnancy test
* Able to communicate well with the investigator, to understand and comply with the requirements of the study
* Signed the written informed consent

Exclusion Criteria:

* Women who are pregnant or lactating or become pregnant during the conduct of the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* Participating in another clinical trial within 30 days
* Malignancy
* Immunosuppression (medication, illness)
* HIV- or Hepatitis infection

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of topical treatment with Imiquimod in patients with CIN 2/3 | 20 weeks after treatment start

SECONDARY OUTCOMES:
HPV-Clearance, feasibility and adverse event profile and drop-out rate | 20 weeks after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Paul Speiser, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Dpt. of General Gynecology and Gynecologic Oncology, Vienna, Austria

REFERENCES:
- [Derived] Grimm C, Polterauer S, Natter C, Rahhal J, Hefler L, Tempfer CB, Heinze G, Stary G, Reinthaller A, Speiser P. Treatment of cervical intraepithelial neoplasia with topical imiquimod: a randomized controlled trial. Obstet Gynecol. 2012 Jul;120(1):152-9. doi: 10.1097/AOG.0b013e31825bc6e8. PMID 22914404